CLINICAL TRIAL: NCT06535503
Title: Clinical Characteristics and Outcomes Among ST-elevation Myocardial Infarction (STEMI) Patients With Cardiogenic Shock at Abu Dhabi City
Brief Title: Clinical Characteristics and Outcomes Among STEMI Patients With Cardiogenic Shock at Abu Dhabi City
Status: Recruiting | Type: Observational
Sponsor: Abu Dhabi Health Services Company (Other Government)
Collaborators: Sheikh Shakhbout Medical City (Other); Sheikh Khalifa Medical City (Other)
Responsible Party: Principal Investigator, Babiker Mohamed Babiker Elsiraj, Principal Investigator, Cardiology Specialist/Fellow at Sheikh Shakhbout Medical City, Abu Dhabi Health Services Company
Other Study IDs: SEHAResearch ID 747
Record Dates: First submitted 2024-05-13; First posted 2024-08-02 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: ST Elevation Myocardial Infarction; Cardiogenic Shock
Keywords: STEMI; Cardiogenic Shock; Morbidity; Mortality
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with STEMI & Cardiogenic Shock: Patients with STEMI complicated by cardiogenic shock on admission or after hospitalization treated at SKMC & SSMC, Abu Dhbai

SUMMARY:
A retrospective study on the clinical characteristics and treatment outcomes of patients admitted with ST-elevation Myocardial Infarction (STEMI) complicated with cardiogenic shock (CS) during admission or CS development during their hospital stay for two tertiary hospitals in Abu Dhabi, UAE, from 2020-2024.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) accounts for 40% of mortality in the UAE, which is higher than the global average. Long-term trends, incidence studies, and best practice guidance on Cardiogenic Shock (CS) with ST-elevation Myocardial infarction (STEMI) in the United Arab Emirates (UAE) and the Gulf Cooperation Council (GCC) are limited.

Through this retrospective study, investigators aim to identify treatment modalities and trends, hospitalization events, and patient demographics and comorbidities which lead to participant recovery or mortality in Sheikh Khalifa Medical City (SKMC) and Sheikh Shakhbout Medical City (SSMC) tertiary hospitals for patients admitted with STEMI and CS or developed CS after hospitalization with STEMI during January 2020-January 2024.[200-400 participants]. Data will be collected from eligible patients' electronic medical records (EMR).

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18.
* STEMI complicated by cardiogenic shock.
* Were hospitalized or treated at SSMC or SKMC for STEMI complicated by cardiogenic shock.
* Patient admitted between January 2019 to March 2024.

Exclusion Criteria:

* Age less than 18.
* Shock patient not related to Myocardial infarction.
* NSTEMI-related cardiogenic shock.
* Patients who were not treated at SSMC or SKMC for the STEMI complicated by cardiogenic shock.
* Patient not admitted between January 2019 to March 2024.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with STEMI complicated by cardiogenic shock on admission or after hospitalization were treated in Abu Dhabi city from January 2020 to January 2024.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Analyze STEMI patient with CS disease profile | 5 years
  Comorbidities, demographical information, past medical history, morbidity
Incidence of CS-complicated AMI events | 5 years
  The incidence of CS-complicated AMI events will show an increase over the years because of advanced diagnostic modalities and a clearer definition of CS.
Analyze treatment outcomes in the targeted population as per the patient profile | 5 years
  Incidence of Mortality
Analyze STEMI patient with CS disease profile | 5 years
  Incidence of Morbidity
Analyze treatment outcomes | 5 years
  % of patients who were discharged

CONTACTS AND LOCATIONS:
Overall Officials: Abdulmajeed BS Alzubaidi, MD, Study Chair — Abu Dhabi Health Services Co. -SEHA; Babiker Babiker Mohamed Babiker Elsiraj MB Elsiraj, Principal Investigator — Sheikh Shakhbout Medical City
Locations (2):
- United Arab Emirates (2):
  - Sheikh Khalifa Medical City (SKMC), Abu Dhabi, Abu Dhabi Emirate
  - Sheikh Shakhbout Medical City (SKMC), Abu Dhabi, Abu Dhabi Emirate

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share the clinical study report with all researchers. We will share the study protocol and case report form if further collaboration is decided while expanding our study.
Supporting Information: CSR
Time Frame: The data will be available for 5 years after the analysis is completed
Access Criteria: REDCap or PI & Facility Permission

REFERENCES:
- [Background] Al-Shamsi S, Regmi D, Govender RD. Incidence of cardiovascular disease and its associated risk factors in at-risk men and women in the United Arab Emirates: a 9-year retrospective cohort study. BMC Cardiovasc Disord. 2019 Jun 17;19(1):148. doi: 10.1186/s12872-019-1131-2. PMID 31208354
- [Background] Akbar H, Mountfort S. Acute ST-Segment Elevation Myocardial Infarction (STEMI). 2024 Oct 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK532281/ PMID 30335314
- [Background] De Luca L, Olivari Z, Farina A, Gonzini L, Lucci D, Di Chiara A, Casella G, Chiarella F, Boccanelli A, Di Pasquale G, De Servi S, Bovenzi FM, Gulizia MM, Savonitto S. Temporal trends in the epidemiology, management, and outcome of patients with cardiogenic shock complicating acute coronary syndromes. Eur J Heart Fail. 2015 Nov;17(11):1124-32. doi: 10.1002/ejhf.339. Epub 2015 Sep 4. PMID 26339723
- [Background] Holmes DR Jr, Bates ER, Kleiman NS, Sadowski Z, Horgan JH, Morris DC, Califf RM, Berger PB, Topol EJ. Contemporary reperfusion therapy for cardiogenic shock: the GUSTO-I trial experience. The GUSTO-I Investigators. Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries. J Am Coll Cardiol. 1995 Sep;26(3):668-74. doi: 10.1016/0735-1097(95)00215-p. PMID 7642857
- [Background] Shalaby G, Niazi AK, Khaled S. Cardiogenic Shock Among Patients with Acute ST-Segment Elevation Myocardial Infarction in a Middle Eastern Country: A Single-Center Experience. J Saudi Heart Assoc. 2023 Jan 20;34(4):232-240. doi: 10.37616/2212-5043.1323. eCollection 2022. PMID 36816794
- [Background] Yusufali A, Bazargani N, Muhammed K, Gabroun A, AlMazrooei A, Agrawal A, Al-Mulla A, Hajat C, Baslaib F, Philip J, Gupta P, Bakir S, Krishnan S, Almahmeed W, Alsheikh-Ali A. Opportunistic Screening for CVD Risk Factors: The Dubai Shopping for Cardiovascular Risk Study (DISCOVERY). Glob Heart. 2015 Dec;10(4):265-72. doi: 10.1016/j.gheart.2015.04.008. Epub 2015 Aug 11. PMID 26271552
- See also: Kosaraju, A., Pendela, V. S., & Hai, O. (2023, April 7). Cardiogenic shock. StatPearls [Internet]. https://www.ncbi.nlm.nih.gov/books/NBK482255/ — https://www.ncbi.nlm.nih.gov/books/NBK482255/
- See also: High prevalence of cardiometabolic risk factors amongst young adults in the United Arab Emirates: The UAE Healthy Future Study. — https://bmccardiovascdisord.biomedcentral.com/articles/10.1186/s12872-023-03165-3